CLINICAL TRIAL: NCT06552416
Title: A Phase 1 Study of Allogenic Off-the-Shelf Multi-Tumor-Associated Antigen-Specific T Cell Products (MT-401-OTS) Administered to Patients With Relapsed Acute Myeloid Leukemia or Myelodysplastic Syndromes (RAPID)
Brief Title: Safety of MT-401-OTS in Patients With Relapsed AML or MDS
Acronym: RAPID
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Marker Therapeutics, Inc. (Industry)
Collaborators: University of Kansas Medical Center (Other); H. Lee Moffitt Cancer Center and Research Institute (Other); City of Hope National Medical Center (Other); FDA Office of Orphan Products Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MRKR-21-401-OTS; 5R01FD007272-02 (FDA)
Record Dates: First submitted 2024-08-07; First posted 2024-08-14 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia, in Relapse; MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: Dose Escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort -1 (Experimental): 50 × 106 cells flat dose, 1 dose infused on Day 0
  Interventions: Drug: MT-401-OTS
- Cohort 1 (Experimental): 100 × 106 cells flat dose, 1 dose infused on Day 0
  Interventions: Drug: MT-401-OTS
- Cohort 2 (Experimental): 200 × 106 cells flat dose, 1 dose infused on Day 0
  Interventions: Drug: MT-401-OTS
- Cohort 3 (Experimental): 400 × 106 cells flat dose, 1 dose infused on Day 0
  Interventions: Drug: MT-401-OTS
- Cohort 4 (optional) (Experimental): up to 400 × 106 cells flat dose TBD based on data from Cohorts 1-3; may include split dosing, dosing with or without lymphodepleting conditioning regimen, or dosing with or without HMA
  Interventions: Drug: MT-401-OTS

INTERVENTIONS:
Drug: MT-401-OTS — MT-401-OTS is an off the shelf cellular therapy product given by IV infusion through either a peripheral or central line.

SUMMARY:
This study is a Phase 1 multicenter, open-label study evaluating the safety and efficacy of escalating doses of MT-401-OTS in 2 participant populations: 1) Those with intermediate or high-risk AML per 2022 ELN criteria who have evidence of MRD and/or </= 10% blast following prior induction therapy or at least 4 cycles of nonintensive therapy and 2) those with high- or very-high-risk MDS per 2023 IWG criteria and who have residual disease with </= 10% blasts following treatment with an HMA-based therapy.

DETAILED DESCRIPTION:
This study is a Phase 1 multicenter, open-label study evaluating the safety and efficacy of escalating doses of MT-401-OTS in 2 participant populations: 1) Those with intermediate or high-risk AML per 2022 ELN criteria who have evidence of MRD and/or </= 10% blast following prior induction therapy or at least 4 cycles of nonintensive therapy and 2) those with high- or very-high-risk MDS per 2023 IWG criteria and who have residual disease with </= 10% blasts following treatment with an HMA-based therapy. Participants must meet all eligibility criteria. Once a suitable MT-401-OTS product is confirmed, the participant will receive a lymphodepleting conditioning regimen consisting of fludarabine and cyclophosphamide daily from Day -7 to Day -5. Bendamustine (administered on Days -6 and -5) may be used for participants with underlying toxicities or if lack of availability precludes the use of fludarabine and/or cyclophosphamide. Two standard doses of an HMA (azacitidine or decitabine) will be administered on Day -4 to -3. MT-401-OTS will be administered IV over 10 minutes on Day 0. Safety evaluations will be performed throughout the study. Disease assessments will be performed at regular intervals based on 2022 ELN criteria for AML and the 2023 response criteria for higher-risk MDS. The dose escalations will begin with Cohort 1 which a single MT-401-OTS dose administered at a flat dose of 100 X 10^6 cells). Dose escalations will proceed using the modified 3+3 design up to the highest single flat dose of 400 x 10^6 cells. If a clinical safety issue should arise in Cohort 1, a lower DL may be explored. Additionally, Cohort 4 is an optional cohort that may be considered based on the cumulative data from Cohorts 1 through 3 to asses alternative dosing schedules (split dosing) of 400 X 10^ 6 cells or without lymphodepletion and/or HMA.

ELIGIBILITY:
Inclusion Criteria:

* General

  1. Must be ≥ 65 years of age and capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in the protocol, at the time of signing the ICF
  2. Must have a life expectancy ≥ 12 weeks
  3. Must have an ECOG performance status of 0-2
  4. Must have available MT-401-OTS product with a ≥ 2/8 HLA match Disease Characteristics
  5. For participants with AML:

     1. Must have a confirmed diagnosis of AML or MDS/AML per 2022 WHO Classification of Haematolymphoid Tumours: Myeloid and Histiocytic/Dendritic Neoplasms or 2022 International Consensus Criteria
     2. Must have intermediate or high-risk disease based on ELN 2022 criteria.
     3. If no targetable mutation is present, must have received 1 prior standard regimen with at least 4 cycles of standard therapy containing an HMA or a standard cytarabine-containing induction therapy
     4. If targetable mutation is present, must have received a regimen that includes commercially available targeted therapy unless unable to tolerate or the participant declines (must be documented in the informed consent). If targeted therapy was not administered as part of first-line of therapy, a second regimen is allowed.
     5. Must have either: ≤ 10% bone marrow blasts and ≤ 5% peripheral blasts during screening and not be considered to have hyperproliferating disease at diagnosis or after treatment OR Evidence of MRD based on evaluation at a local laboratory
  6. For participants with MDS:

     1. Must have confirmed diagnosis of MDS based on 2022 WHO Classification of Haematolymphoid Tumours: Myeloid and Histiocytic/Dendritic Neoplasms or 2022 ICC criteria
     2. Must have high-risk or very-high-risk disease based on IPSS-M (ie, not evolved to AML)
     3. Must have received standard treatment with at least 4 cycles of an HMA and have evidence of continued disease, including morphologic disease or MRD-positive
     4. Must have bone marrow blasts ≤ 10% at screening Health Status
  7. Must have adequate coagulation, hepatic, renal, and cardiac function:

     1. PT/INR and PTT/aPTT < 1.3 × ULN
     2. AST and ALT < 3 × ULN; for participants with leukemic infiltration of the liver (documented by biopsy or imaging), AST and ALT < 5 × ULN is permitted.
     3. Total bilirubin ≤ 1.5 × ULN unless bilirubin rise is due to Gilbert's syndrome or of nonhepatic origin (2 × ULN is permitted)
     4. eGFR ≥ 40 mL/min by the MDRD formula
     5. LVEF ≥ 45% (prior to apheresis and lymphodepletion) Sex
  8. Women of childbearing potential are eligible to participate if they agree to the following during the intervention period and for at least 1 year after the last infusion of MT-401-OTS:

     1. Must use a contraceptive method that is highly effective (ie, with a failure rate of < 1% per year; see Section 10.3), preferably with low user dependency PLUS
     2. Must agree not to donate eggs (ie, ova and oocytes) for the purpose of reproduction
  9. Male participants are eligible to participate if they agree to the following during the intervention period and for at least 6 months after the last infusion of MT-401-OTS:

     1. Must refrain from donating sperm

        PLUS either:
     2. Must be abstinent from intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent OR
     3. Must agree to use a male condom AND should also be advised of the benefit for a nonpregnant female partner to use a highly effective method of contraception (see Section 10.3) as a condom may break or leak

Exclusion Criteria:

* Disease-Related

  1. Have leukemic involvement in the CNS
  2. Have other extramedullary disease involvement (except hepatosplenic involvement)
  3. Have APL Medical Conditions
  4. Have primary immunodeficiency
  5. Have severe or uncontrolled autoimmune disorder
  6. Have a history or presence of clinically relevant CNS pathology, such as epilepsy, seizure, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome or psychosis
  7. Have active malignancies (ie, those that are progressing or have required treatment change in the last 24 months) other than the disease being treated under study. Exceptions to this inclusion include the following:

     1. Nonmelanoma skin cancer treated within the last 24 months that is considered completely cured
     2. Adequately treated breast lobular carcinoma in situ and breast ductal carcinoma in situ
     3. Adequately treated cervical carcinoma in situ without evidence of disease
     4. History of localized breast cancer and receiving antihormonal agents, or history of localized prostate cancer (N0M0) and receiving androgen-deprivation therapy
     5. A malignancy that is considered cured with minimal risk of recurrence
  8. Have any active systemic infection requiring therapy (viral, bacterial, or fungal), including HIV
  9. Have active hepatitis B or C infection or other clinically active liver diseases, as defined below:

     1. Seropositivity for hepatitis B as defined by a positive test for HbsAg Participants with resolved infection (ie, participants who are HbsAg-negative with antibodies to total anti-HBc with or without the presence of anti-HBs) must be screened using RT-PCR measurement of HBV DNA levels. Those who are RT PCR-positive will be excluded.

        Participants with serologic findings suggestive of HBV vaccination (anti HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by RT PCR.
     2. Active hepatitis C infection as defined by being positive for a nucleic acid test for HCV RNA
  10. Have Class III or IV congestive heart failure per New York Association
  11. Have unstable angina
  12. Have a history or evidence of current, uncontrolled, clinically significant, unstable arrhythmias
  13. Have an oxygen saturation on room air of ≤ 92%
  14. Have clinically significant reversible nonhematologic toxicities from prior cancer therapy that have not recovered to Grade 1 or baseline Note: Participants with clinically nonsignificant toxicities, such as asymptomatic laboratory values, will be allowed on study.

      Prior/Concomitant Therapies
  15. Received prior treatments for underlying malignancy, except as specified in the Inclusion Criteria. Participants with AML secondary to MDS may have received prior treatment for MDS.
  16. Have had prior HSCT
  17. Are receiving concurrent therapies other than HMA, as delineated in the study design
  18. Have received hematopoietic growth factors within 2 days of lymphodepleting conditioning regimen
  19. Have a history of severe allergic reactions/intolerance to any of the study intervention components, including the conditioning regimen, HMA, or DSMO, or to tocilizumab
  20. Have had major surgery within 14 days (central line placement allowed)
  21. Have received systemic steroids (exception: physiological doses of steroids allowed) or other immunosuppressive therapies within 14 days prior to lymphodepleting conditioning regimen Other
  22. Are unable to be matched with MT-401-OTS product inventory
  23. Are pregnant or breastfeeding
  24. Have any other issue that, in the opinion of the treating physician, would make the participant ineligible for the study or unable to comply with its requirements

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Safety of MT-401-OTS | Through study completion. Approximately 5 years
  Assess:
  * Incidence of DLTs to determine the RP2D
  * Safety (including but not limited to): TEAEs, SAEs, deaths, and clinical laboratory abnormalities per NCI CTCAE, Version 5.0
  * Acute GVHD per 2016 MAGIC criteria
  * CRS and ICANS per ASTCT criteria
Tolerability of MT-401-OTS | Through study completion. Approximately 5 years
  cGVHD per 2014 NIH consensus criteria for cGVHD

SECONDARY OUTCOMES:
To assess the efficacy of MT-401-OTS in participants with high-risk or very-high-risk MDS per IPSS-M who have evidence of disease following at least 4 cycles of a HMA | Following conclusion of the disease assessment of last MDS subject treated. Approximately 2 years
  Per 2023 IWG criteria for higher-risk MDS:
  * CR rate
  * DOCR
  * ORR
  * DOR
To assess the efficacy of MT-401-OTS in participants with intermediate or high-risk AML per 2022 ELN criteria who have evidence of disease following induction therapy or at least 4 cycles of nonintensive treatment | Following conclusion of the disease assessment of last AML subject treated. Approximately 2 years
  Per 2022 ELN Criteria for AML:
  * Rate of MRD negativity
  * CR, DOCR
  * ORR, DOR

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - City of Hope Center (City of Hope National Medical Center, City of Hope Medical Center), Duarte, California
  - Moffitt Cancer Center, Tampa, Florida
  - KU Cancer Center, Kansas City, Kansas

IPD SHARING:
Plan to Share IPD: No
IPD sharing plan will be developed once it is determined that the results of this study may be published or presented at scientific meetings.